CLINICAL TRIAL: NCT02545855
Title: Long-term High-flow Nasal Cannula Therapy in Patients With Stable COPD: a Prospective, Randomized Crossover Study
Brief Title: High-flow Nasal Cannula Therapy for Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Kobe City Medical Center General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TRIRES1507; UMIN000017639 (Other: UMIN-CTR)
Record Dates: First submitted 2015-09-01; First posted 2015-09-10 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: myAIRVO2; high-flow nasal cannula therapy; home oxygen therapy; HOT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (myAIRVO2® + HOT, HOT) (Experimental): Subjects will receive the myAIRVO2® therapy plus HOT for week 1-6 and HOT only for week 7-12. After treatment period (week 1-12), willing subjects can continue the myAIRVO2® therapy plus HOT for week 13-52 regardless of treatment arm assignment.
  Interventions: Device: High-flow nasal cannula therapy; Device: Home oxygen therapy (HOT)
- Arm B (HOT, myAIRVO2® + HOT) (Experimental): Subjects will receive HOT only for week 1-6 and the myAIRVO2® therapy plus HOT for week 7-12. After treatment period (week 1-12), willing subjects can continue the myAIRVO2® therapy plus HOT for week 13-52 regardless of treatment arm assignment.
  Interventions: Device: High-flow nasal cannula therapy; Device: Home oxygen therapy (HOT)

INTERVENTIONS:
Device: High-flow nasal cannula therapy — All subjects will receive nocturnal high-flow nasal cannula therapy with the myAIRVO2®, in addition to their current HOT. The myAIRVO2® is used for at least 4 hours per day with flow rates in the range 30-40 L/min. The investigator can adjust the nocturnal oxygen flow rates to keep SpO2 88-92% stably. If the subjects report discomfort, the investigator can adjust the flow rates in the range at least 20 L/min.
  Other Names: myAIRVO2®
Device: Home oxygen therapy (HOT) — All subjects will continue their current HOT which kept original usage conditions at the time of enrollment throughout the entire duration of the study regardless of treatment arm assignment.

SUMMARY:
This is a prospective, randomized crossover study for evaluation of the efficacy and safety of long-term nocturnal high-flow nasal cannula therapy with the myAIRVO2® in stable COPD patients with stage 2-4 of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) and hypercapnia who require home oxygen therapy (HOT). The total duration of subject participation will be 52 weeks, consisting of 12-week treatment period and 40-week continuation period. Subjects who satisfy all inclusion and exclusion criteria will be randomly assigned to one of two treatment arms, Arm A (week 1-6: the myAIRVO2® therapy plus HOT, week 7-12: HOT only) or Arm B (week 1-6: HOT only, week 7-12: the myAIRVO2® therapy plus HOT). All subjects will receive nocturnal high-flow nasal cannula therapy with the myAIRVO2®, in addition to their current HOT. After treatment period, the willing subjects can continue the myAIRVO2® therapy plus HOT for week 13-52 regardless of treatment arm assignment. The end of the study is defined as the treatment period or continuation period end date of the last participant, whichever is later. Subjects will primarily be assessed by the St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at week 0, 6, 12, 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with the Global Initiative for Obstructive Lung Disease (GOLD) stage 2-4 COPD
2. Subjects who have received HOT for at least 16 hours per day for at least 1 month at the time of informed consent
3. Subjects with PaCO2 <= 60 torr, and >= 45 torr at the time of screening
4. Subjects who have signed written informed consent to participate in this study

Exclusion Criteria:

1. Subjects with severe kidney, liver or cardiovascular disease
2. Subjects with active malignant tumor
3. Subjects with acute disease (i.e., acute myocardial infarction)
4. Subjects with a history of obstructive sleep apnea syndrome
5. Subjects with complications affecting efficacy endpoints and who are regarded by the investigator as inadequate for this study
6. Subjects who had experienced COPD exacerbation within the past 6 weeks prior to informed consent
7. Subjects who have been receiving nocturnal noninvasive positive pressure ventilation (NPPV) or had been received within the past 6 weeks prior to informed consent
8. Subjects with a history of tracheotomy or severe pharyngeal nasal cavity surgery within the past 6 months
9. Pregnant women
10. Subjects with cognitive impairment or mental disorder and who are regarded by the investigator as inadequate to be evaluated in this study
11. Subjects who are regarded by the investigator as being unable to operate the myAIRVO2 adequately at home
12. Subjects who are participating or wil participate in the another clinical trial at the time of informed consent
13. Any other cases who are regarded by the investigator as inadequate for enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08-17 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the St. George's Respiratory Questionnaire for COPD patients (SGRQ-C) total score at week 6 and 12 | Week 0, 6 and 12

SECONDARY OUTCOMES:
Quality-adjusted life year (QALY) by Japanese version of the EQ-5D-5L value sets | Week 0, 6, 12 and 52
  Quality-adjusted life year (QALY) of subjects will be assessed by Japanese version of the EQ-5D-5L value sets at week 6 and 12, including assessment of changes from baseline in the EQ-5D-5L utility index scores and visual analogue scale scores at week 6, 12 and 52.
Changes from baseline in symptom, activity and impact scores of the St. George's respiratory questionnaire for COPD patients (SGRQ-C) at week 6 and 12 | Week 0, 6 and 12
Changes from baseline in the modified medical research council (mMRC) scale at week 6 and 12 | Week 0, 6 and 12
Changes from baseline in potential hydrogen (pH), partial pressure of oxygen (PaO2), and partial pressure of carbon dioxide (PaCO2) of the arterial blood gas analysis at week 6 and 12 | Week 0, 6 and 12
Changes from baseline in oxygen saturation (SpO2) at week 6 and 12 | Week 0, 6 and 12
Changes from baseline in transcutaneous carbon dioxide (PtcCO2) levels and the median - 95th percentile of nocturnal transcutaneous carbon dioxide (PtcCO2) at week 6 and 12 | Week 0, 6 and 12
Changes from baseline in the pulmonary function tests at week 6 and 12 | Week 0, 6 and 12
  Lung function of subjects will be assessed by the pulmonary function tests in the following indicators: vital capacity (VC, %VC), forced vital capacity (FVC, %FVC), forced expiratory volume in 1 second (FEV1, ％FEV1), FEV1/FVC, diffusion capacity to carbon monoxide (DLCO, %DLCO), residual volume (RV, %RV), functional residual capacity (FRC, %FRC) and total lung capacity (TLC, %TLC).
Changes from baseline in the 6-minute walk test (6MWT) scores at week 6 and 12 | Week 0, 6 and 12
  Functional exercise capacity of subjects will be assessed by the 6MWT in the following indicators: the 6MWT distance (m), changes in pre- and post-6MWT pulse oximeter (SpO2), and post-6MWT modified borg scale.
Changes from baseline in physical activity by the Lifecorder® at week 6 and 12 | Week 0, 6 and 12
  Physical activity of subjects will be assessed by the Lifecorder® in the daily average of the following indicators: energy consumption (kcal/day), step-counts (steps/d) and activity time (h/d). The indicators will be calculated by 7 days records just before each assessment day.
COPD exacerbation in both week 1-6 and week 7-12 | Week 1-6 and week 7-12
Medication change | Week 1-52
Oxygen flow rate at pre- and post-myAIRVO2® therapy in treatment period (week 1-12) | Week 1-12
Total flow rates at pre- and post-myAIRVO2® therapy in treatment period (week 1-12) | Week 1-12
Hours of receiving the myAIRVO2® therapy in treatment period (week 1-12) | Week 1-12
Adverse events with an undeniable causal relationship to the myAIRVO2® therapy | Week 1-52

OTHER OUTCOMES:
The ratio of subjects received the myAIRVO2® therapy plus HOT at least 1 day in continuation period (week 13-52) in subjects who completed treatment period (week 1-12) | Week 13-52
Duration from initial date of continuation period (week 13-52) until the date of first COPD exacerbation | Week 13-52
Chronological changes of symptom, activity and impact scores of the St. George's respiratory questionnaire for COPD patients (SGRQ-C) in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52
Chronological changes of the modified medical research council (mMRC) scale in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52
Chronological changes of potential hydrogen (pH), partial pressure of oxygen (PaO2), and partial pressure of carbon dioxide (PaCO2) of the arterial blood gas analysis in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52
Chronological changes of oxygen saturation (SpO2) in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52
Chronological changes of transcutaneous carbon dioxide (PtcCO2) levels and the median - 95th percentile of nocturnal transcutaneous carbon dioxide (PtcCO2) in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52
Chronological changes of the pulmonary function tests in subjects having a full data set at week 0, 6, 12, 24 and 52 | Week 0, 6, 12, 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Tomii, MD, Ph.D., Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan

REFERENCES:
- [Derived] Nagata K, Kikuchi T, Horie T, Shiraki A, Kitajima T, Kadowaki T, Tokioka F, Chohnabayashi N, Watanabe A, Sato S, Tomii K. Domiciliary High-Flow Nasal Cannula Oxygen Therapy for Patients with Stable Hypercapnic Chronic Obstructive Pulmonary Disease. A Multicenter Randomized Crossover Trial. Ann Am Thorac Soc. 2018 Apr;15(4):432-439. doi: 10.1513/AnnalsATS.201706-425OC. PMID 29283682